CLINICAL TRIAL: NCT07215988
Title: Studying Off Label Insurance Coverage for Patients With Cutaneous Cancers a "Filter" Observational Study
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Claire Verschraegen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-23272; NCI-2025-07206 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Clinical Stage II Cutaneous Merkel Cell Carcinoma AJCC v8; Clinical Stage III Cutaneous Merkel Cell Carcinoma AJCC v8; Clinical Stage IV Cutaneous Merkel Cell Carcinoma AJCC v8; Locally Advanced Basal Cell Carcinoma; Locally Advanced Malignant Skin Neoplasm; Locally Advanced Merkel Cell Carcinoma; Locally Advanced Mucosal Melanoma; Locally Advanced Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Cohort 1: Merkel cell carcinoma: Patients complete a survey and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study
- Cohort 2: Mucosal melanoma: Patients complete a survey and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study
- Cohort 3: Basal cell carcinoma: Patients complete a survey and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study
- Cohort 4: Rare cutaneous cancers: Patients complete a survey and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study evaluates the time spent on obtaining insurance approval and drugs, means of insurance coverage, out-of-pocket costs for patients, and the surgical outcomes after neoadjuvant treatment is completed in skin cancer patients receiving "off label" and "on label" neoadjuvant treatment. "Neoadjuvant therapy" means cancer treatment given before surgery. However, in many instances, neoadjuvant therapy is used as an "off-label" approach for several types of skin cancers. "Off-label" means that the FDA has not yet approved its use for that type of cancer. Therefore, insurance approval of these "off-label" treatments could be delayed compared to label use, and "off-label" treatments may require several weeks of pre-authorization. There is evidence that the delayed start of cancer treatment can lead to poorer outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess in real-life clinical practice, the timing, cost, and surgical outcomes of patients who have resectable various skin cancers that are locally advanced or have a high risk of recurrence.

OUTLINE: This is an observational study.

Patients complete a survey and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* * MERKEL CELL CARCINOMA

  * Signed informed consent
  * Pathology report confirming Merkel at the time of screening
  * Stage II, III or IV resectable (criteria based on Merkel Cell carcinoma TNM pathologic staging AJCC UICC 8th edition) or unresectable cancers amenable to surgery if a response is elicited with neoadjuvant therapy
  * ≥ 18 years of age
  * Genomics of the cancer attempted
  * Description of planned surgical resection by surgeon
  * Planned treatment with immunotherapy. Possible Beacon plan entitled OP NIVOLUMAB IPILIMUMAB NEUROENDOCRINE (PRL 8149)

    * 2 cycles will be given prior to surgery (=12 weeks).

      * MUCOSAL MELANOMA
  * Signed informed consent
  * Pathology report confirming mucosal melanoma at the time of screening
  * Stage III or IV resectable (TNM pathologic staging AJCC UICC 8th edition) or unresectable cancers amenable to surgery if a response is elicited with neoadjuvant therapy
  * ≥ 18 years of age
  * Genomics of the cancer attempted
  * Description of planned surgical resection by surgeon
  * SOC (standard of care) treatment planned with immunotherapy Possible Beacon plan entitled OP NIVOLUMAB IPILIMUMAB -> NIVOLUMAB Q4 WEEK MAINTENANCE MELANOMA 4 cycles will be given prior to surgery (=12 weeks)

    * BASAL CELL CARCINOMA
  * Signed informed consent
  * Pathology report confirming basal cell carcinoma with subtype at the time of screening
  * Resectable tumor of any stage, or unresectable tumor that could be amenable to surgery if there is a good response.
  * ≥ 18 years of age
  * Genomics of the cancer attempted
  * Description of planned surgical resection by surgeon
  * SOC treatment planned with possible Beacon plan entitled OP SONIDEGIB BASAL CELL CARCINOMA 3 months will be given prior to surgery (= 12 weeks) (Vismodegib may be substituted if current national shortage of sonidegib persists)

    * RARE CUTANEOUS CANCERS
  * Signed informed consent
  * Pathology report confirming squamous cell carcinoma at the time of screening
  * Stage II, III, or IV resectable or (TNM pathologic staging AJCC UICC 8th edition) or unresectable cancers amenable to surgery if a response is elicited with neoadjuvant therapy
  * ≥ 18 years of age
  * Genomics of the cancer attempted
  * Description of planned surgical resection by surgeon
  * Planned SOC treatment with possible Beacon plan entitled OP WEEKLY CARBOPLATIN PACLITAXEL + PEMBROLIZUMAB Q3 WEEKS HEAD AND NECK

    * 4 cycles will be given prior to surgery (= 12 weeks)

Exclusion Criteria:

* * MERKEL CELL CARCINOMA

  * Metastatic disease not amenable to complete resection
  * Prior immunotherapy, chemotherapy, or radiation therapy for treatment of MCC
  * Any clinically significant medical condition, which in the judgment of the attending physician would contraindicate immunotherapy
  * Is pregnant or breast feeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of SOC treatment.

    * MUCOSAL MELANOMA
  * Metastatic disease not amenable to complete resection
  * Prior immunotherapy, chemotherapy, or radiation therapy for treatment of this mucosal melanoma
  * Any clinically significant medical condition, which in the judgment of the attending physician would contraindicate immunotherapy
  * Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of SOC treatment.

    * BASAL CELL CARCINOMA
  * Metastatic disease not amenable to complete resection
  * Prior immunotherapy, chemotherapy, or radiation therapy for treatment of this basal cell carcinoma
  * Any clinically significant medical condition, which in the judgment of the attending physician would contraindicate immunotherapy
  * Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of SOC treatment.

    * RARE CUTANEOUS CANCERS
  * Metastatic disease not amenable to complete resection
  * Prior immunotherapy, chemotherapy, or radiation therapy for treatment of this mucosal melanoma
  * Any clinically significant medical condition, which in the judgment of the attending physician would contraindicate immunotherapy
  * Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of SOC treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Merkel cell carcinoma, mucosal melanoma, basal cell carcinoma, and miscellaneous rare cutaneous cancers will be recruited from The James Comprehensive Cancer Center during the course of usual care.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time spent obtaining approval and drugs | Up to study completion, up to 17 weeks
  Start and end times for obtaining approval for drugs will be based on date the initial request is submitted by the provider and the date the drugs are obtained. Confidence intervals will provide precision for estimating the mean time spent on obtaining approval and drugs and out-of-pocket expenses for patients.
Means of coverage | Up to study completion, up to 17 weeks
  Descriptive statistics will summarize the conditions of off label coverage among patients, with mean, median, interquartile range, min, and max for continuous variables and frequencies / percentages for categorical variables.
Out of pocket expenses for patients | Up to study completion, up to 17 weeks
  Descriptive statistics will summarize the conditions of off label coverage among patients, with mean, median, interquartile range, min, and max for continuous variables and frequencies / percentages for categorical variables.
Extent of surgical resection | Up to study completion, up to 17 weeks
  Planned vs empirical extent of surgical resection will be calculated and compared within each cohort, with Clopper-Pearson exact binomial 95% confidence intervals for the percent of patients receiving lesser extent of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Claire F Verschraegen, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu